CLINICAL TRIAL: NCT03653832
Title: Alpha 2 Agonists for Sedation to Produce Better Outcomes From Critical Illness (A2B Trial): A Randomised, Parallel-group, Allocation Concealed, Controlled, Open, Phase 3 Pragmatic Clinical and Cost- Effectiveness Trial With Internal Pilot
Brief Title: Alpha 2 Agonists for Sedation to Produce Better Outcomes From Critical Illness (A2B Trial)
Acronym: A2B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: West Hertfordshire Hospitals NHS Trust (Other); Queen's University, Belfast (Other); The University of Queensland (Other); University Hospital of Wales (Other); Edinburgh Napier University (Other); King's College London (Other); University of Warwick (Other); University of Manchester (Other); Royal Surrey County Hospital NHS Foundation Trust (Other); University College, London (Other); NHS Lothian (Other Government); Imperial College London (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC18022; HTA 16/93/01 (Other Grant/Funding Number: NIHR HTA Programme); 2018-001650-98 (EudraCT Number); 243640 (Other: Integrated Research Application System (IRAS)); 18/SS/0085 (Other: REC Number)
Record Dates: First submitted 2018-08-21; First posted 2018-08-31 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Critical Illness
Keywords: Sedation; Ventilation
MeSH Terms: conditions — Critical Illness; Respiratory Aspiration | interventions — Dexmedetomidine; Clonidine; Propofol

STUDY DESIGN:
Intervention Model Description: A randomised, parallel-group, allocation concealed, controlled, open, phase 3 pragmatic clinical and cost- effectiveness trial with internal pilot
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine Group (Experimental): For dexmedetomidine, the regimen will follow the manufacturer's guidance and regimens used in previous trials. Dexmedetomidine will be up and down titrated against sedation targets set by clinical staff and reviewed at regular intervals, and documented at least daily. No loading dose will be administered. The starting dose will be 0.7 µg.kg-1.hour-1 titrated to a maximum dose 1.4 µg.kg-1 hour-1. Lower starting doses will be used at clinical discretion for patients with cardiovascular instability.
  Interventions: Drug: Dexmedetomidine
- Clonidine Group (Experimental): For clonidine, the regimen is designed to be equipotent with dexmedetomidine based on known pharmacokinetics and pharmacodynamics. The chosen regimen is similar to that currently used in many UK ICUs as part of routine 'off label' practice. Clonidine will be up and down titrated against sedation targets set by clinical staff and reviewed at regular intervals, and at least daily. No loading dose will be administered. The starting dose will be 1.0µg.kg-1.hour-1 titrated to a maximum dose of 2 µg.kg-1.hour-1. Lower starting doses will be used at clinical discretion for patients with cardiovascular instability.
  Interventions: Drug: Clonidine
- Usual Care (Propofol) Group (Active Comparator): Usual Care Group : Patients will continue to receive intravenous propofol according to usual current care . The sedation targets, weaning, and sedation discontinuation procedures will follow the same clinical targets as for the clonidine and dexmedetomidine groups.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will commence intravenous infusion of open-label study drug according to a weight-based dose regimen as early as possible post-randomisation, and within a maximum of two hours.
  Bedside clinical staff will transition patients to achieve sedation with the allocated α2-agonist agent as quickly as clinically feasible and safe, to replicate the way these drugs would be used in routine practice. Additional opiate will be used for analgesia using clinical judgement. Once established, additional propofol will only be used when the maximum α2-agonist dose is reached or because cardiovascular or other side-effects limit dose escalation.
  Other Names: Dexdor
  Arms: Dexmedetomidine Group
Drug: Clonidine — Patients will commence intravenous infusion of open-label study drug according to a weight-based dose regimen as early as possible post-randomisation, and within a maximum of two hours.
  Bedside clinical staff will transition patients to achieve sedation with the allocated α2-agonist agent as quickly as clinically feasible and safe, to replicate the way these drugs would be used in routine practice. Additional opiate will be used for analgesia using clinical judgement. Once established, additional propofol will only be used when the maximum α2-agonist dose is reached or because cardiovascular or other side-effects limit dose escalation.
  Other Names: Catapres
  Arms: Clonidine Group
Drug: Propofol — Patients will continue to receive intravenous propofol according to current usual care.
  Other Names: Diprivan
  Arms: Usual Care (Propofol) Group

SUMMARY:
Many patients in intensive care (ICU) need help to breathe on a breathing machine and need pain killers and sedatives to keep them comfortable and pain free. However, keeping patients too deeply sedated can make their ICU stay longer, can cause ICU confusion (delirium) and afterwards may cause distressing memories. Ideally patients should be kept less sedated, but it is difficult to get the balance of sedation and comfort right.

The investigators want to know whether starting an alpha2-agonist drug early in ICU can help keep patients more lightly sedated but still comfortable, and whether patients spend less time on the ventilator. The investigators also want to know how safe they are and if they can improve important outcomes during ICU stay and during recovery. The investigators also want to know if they are value for money.

DETAILED DESCRIPTION:
Many patients in intensive care (ICU) need help to breathe on a breathing machine and need pain killers and sedatives to keep them comfortable and pain free. However, keeping patients too deeply sedated can make their ICU stay longer, can cause ICU confusion (delirium), and afterwards may cause distressing memories. Ideally, the investigators want to keep patients less sedated, but it is difficult to get the balance of sedation and comfort right.

For sedation, most ICUs use a drug called 'propofol' that is good at reducing anxiety and making people sleepy, but is not a pain killer, so additional pain killers are needed. There are two other drugs used less often called 'alpha-2 agonists' that have both sedative and pain-killing actions, which may make it easier for patients to be more awake and comfortable on the ventilator. The two drugs are called clonidine and dexmedetomidine.

The investigators want to know whether starting an alpha2-agonist drug early in ICU, and using this instead of propofol as much as possible, can help keep patients more lightly sedated but still comfortable, and whether patients spend less time on the ventilator with these drugs. The investigators also want to know how safe these drugs are and if improve important outcomes during ICU stay can be improved (like delirium, comfort, and safety) and during recovery (like bad memories, anxiety, and depression). The investigators also want to know if they are value for money.

The trial will include 1437 participants needing to be on a ventilator for at least 2 days. Participants will be allocated to one of three groups by chance. One group will continue to receive propofol; one group will receive dexmedetomidine; and one group will receive clonidine. All participants will receive extra pain relief if needed, and participants in the dexmedetomidine and clonidine groups will continue to receive propofol if they need this in addition. Nurses and doctors will alter the doses of sedation drugs to try and reduce or stop them, but always aiming to have participants lightly sedated and comfortable. The trial will compare if participants on dexmedetomidine or clonidine come off the ventilator quicker than those just on propofol. The trial will examine whether there was a difference between the groups in the number of participants who experienced delirium in ICU, compare how comfortable participants were, and measure if participants memories of being in the ICU differed.

Patients who were in the trial will be followed up for up to 180 days afterwards because the investigators want to compare if there were differences in the after-effects of being ill in ICU between the groups. Participants will be asked to complete questionnaires that will assess their memories of the ICU experience at 90 days after entering the trial. At 180 days, participants will be asked to complete questionnaires so that the investigators can detect how patients feel about their quality of life or if they suffer from anxiety, depression or stress. Note that for patients recruited during the final months of recruitment, the 90 and 180 days follow will be truncated and not collected. This was agreed with the TSC and funder to reduce trial costs and enable trial completion.

Alongside this trial, investigators will be looking at value for money, which is important because clonidine, dexmedetomidine, and propofol costs are quite different. Clonidine, in particular, is relatively inexpensive. ICU nurses' and doctors' views on how easy or difficult it was to adjust and use the drugs will be obtained. This will give valuable practical information that can be shared with other ICUs, particularly if alpha2-agonists are found to be better and other ICUs want to start using them.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring mechanical ventilation (MV) in an ICU
2. Aged 18 or over
3. Within 48 hours of first episode of mechanical ventilation in ICU
4. Requiring sedation with propofol
5. Expected to require a total of 48 hours of MV or more in ICU
6. Expected to require a further 24 hours of MV or more at the time of randomisation in the opinion of the responsible clinician

Exclusion Criteria:

1. Acute brain injury (traumatic brain injury; intracranial haemorrhage; ischaemic brain injury from stroke or hypoperfusion)
2. Post-cardiac arrest (where there is clinical concern about hypoxic brain injury)
3. Status epilepticus
4. Continuous therapeutic neuromuscular paralysis at the time of screening or randomisation
5. Guillain-Barre Syndrome
6. Myasthenia gravis
7. Home ventilation
8. Fulminant hepatic failure
9. Patient not expected to survive 24 hours by responsible clinician
10. Decision to provide only palliative or end-of-life care
11. Pregnancy
12. Known allergy to one of the study drugs
13. Untreated second or third degree heart block
14. Transferred from another Intensive Care Unit in which MV occurred for >6 hours
15. Prisoners
16. Enrolled on another CTIMP
17. Previously enrolled on the A2B Trial
18. Patient known to have experienced a period with heart rate <50 beats per minute for 60 minutes or longer since commencing mechanical ventilation in the ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1437 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Time to first successful extubation post-randomisation (hours). | Ventilation status will be recorded twice daily from the date of randomisation until the date of documented successful extubation, or 180 days, whichever comes first.
  How many hours are participants on the study ventilated for?

SECONDARY OUTCOMES:
Length of ICU stay | ICU status will be recorded daily from the date of randomisation until the date of ICU discharge, or 180 days, whichever comes first.
  Number of days the participant is in ICU
Delirium prior to successful extubation | Delirium will be assessed twice daily during ICU stay using the Confusion-Agitation method for ICU (CAM-ICU). Delirium will be assessed from the date of randomisation until the date of ICU discharge, or 28 days, whichever comes first.
  Did participants have delirium during ICU stay?
Duration of Delirium during ICU stay | Delirium will be assessed twice daily during ICU stay using the Confusion-Agitation method for ICU (CAM-ICU). Delirium will be assessed from the date of randomisation until the date of ICU discharge, or 28 days, whichever comes first.
  How many days did participants have delirium during their ICU stay?
Sedation quality as measured by Richmond Agitation and Sedation Scale (RASS) | Sedation quality will be assessed 4 hourly during the period of ventilation from the date of randomisation until the participant is successfully extubated, or 28 days, whichever comes first.
  Sedation quality as measured by Richmond Agitation and Sedation Scale (RASS). RASS scale ranges from -5 to +4. optimal score is between -2 and +1.
Sedation quality as measured by Sedation Quality Assessment Tool (SQAT) | Sedation quality will be assessed daily during the period of ventilation from the date of randomisation until the participant is successfully extubated, or 28 days, whichever comes first.
  Two components of the SQAT assessment will be used in this trial to measure sedation quality.
Analgesia quality as measured by Richmond Agitation and Sedation Scale (RASS) | Analgesia quality will be assessed 4 hourly during the period of ventilation from the date of randomisation until the participant is successfully extubated, or 28 days, whichever comes first.
  Quality of Analgesia measured by Richmond Agitation and Sedation Scale (RASS). RASS scale ranges from -5 to +4. optimal score is between -2 and +1.
Analgesia quality as measured by Sedation Quality Assessment Tool (SQAT) | Analgesia quality will be assessed daily during the period of ventilation from the date of randomisation until the participant is successfully extubated, or 28 days, whichever comes first.
  Quality of Analgesia measured by Sedation Quality Assessment Tool (SQAT)
Number of hours to first optimum sedation as measured by a RASS score of -2 or greater | Level of sedation will be assessed 4 hourly during the period of ventilation from the date of randomisation until the participant is successfully extubated, or 28 days, whichever comes first.
  Number of hours to first optimum sedation as measured by a RASS score of -2 or greater
Number of days to first optimum sedation as assessed by the Sedation Quality Assessment Tool (SQAT) | Level of sedation will be assessed daily during the period of ventilation from the date of randomisation until the participant is successfully extubated, or 28 days, whichever comes first.
  Number of days to first optimum sedation as assessed by the Sedation Quality Assessment Tool (SQAT)
Ability to communicate pain | Ability to communicate pain will be assessed twice daily during the period of ventilation from the date of randomisation until the participant is successfully extubated, or 28 days, whichever comes first.
  Binary assessment by bedside nurse
Ability to co-operate with care | Ability to co-operate with care will be assessed twice daily during the period of ventilation from the date of randomisation until the participant is successfully extubated, or 28 days, whichever comes first.
  Binary assessment by bedside nurse
Relative/Partner/Friend (PerLR) assessment of wakefulness | Participant wakefulness will be assessed by a Relative/Partner/Friend daily during the period of ventilation from the date of randomisation until the participant is successfully extubated, or 28 days, whichever comes first.
  PerLR response to verbal question
Relative/Partner/Friend (PerLR) assessment of patient comfort | Comfort of participant will be assessed by a Relative/Partner/Friend daily during the period of ventilation from the date of randomisation until the participant is successfully extubated, or 28 days, whichever comes first.
  PerLR response to verbal question
Relative/Partner/Friend (PerLR) assessment of patient communication | Participant communication will be assessed by a Relative/Partner/Friend daily during the period of ventilation from the date of randomisation until the participant is successfully extubated, or 28 days, whichever comes first.
  PerLR response to verbal question
Incidence of Drug-related adverse events - Bradycardia; hypotension; hypertension; cardiac arrhythmias; cardiac arrest | The incidence of drug-related adverse events as documented in the medical records will be recorded daily from the date of randomisation until the date of documented successful extubation, or 28 days, whichever comes first.
  Incidence of drug-related adverse events as documented in the medical records
Incidence of Mortality | The incidence of death as documented in the medical records will be recorded from the date of randomisation until the date of the last follow-up visit at 180 days.
  Mortality data collected from medical records
Patient experience of ICU care measured at 90 days | 90 days post ICU discharge
  Patient experience of ICU care measured by Intensive Care Experience Questionnaire
Occurrence of Anxiety and depression at 180 days | 180 days post ICU discharge
  Patient anxiety and depression measured by Hospital Anxiety and Depression Scale (HADS) questionnaire
Occurrence of Post-traumatic stress at 180 days | 180 post ICU discharge
  Occurence of post-traumatic stress measured by Impact of Events Scale-revised (IES-R)
Cognitive function assessed at 180 days using the Montreal Cognitive Assessment Tool (Postal or Telephone) | 180 days post ICU discharge
  Cognitive function assessed at 180 days using the Montreal Cognitive Assessment Tool (Postal or Telephone)
Health related Quality of Life (recalled) assessed by Euroqol tool (EQ-5D-5L) | 30 days post ICU discharge - recalled prior to hospital admission
  Health related Quality of Life (recalled) assessed by Euroqol tool (EQ-5D-5L). Scale is between 5-25 which lower scores having the better outcome.
Health related Quality of Life (30 day) assessed by Euroqol tool (EQ-5D-5L) | 30 days post ICU discharge
  Health related Quality of Life (30 day) assessed by Euroqol tool (EQ-5D-5L). Scale is between 5-25 which lower scores having the better outcome.
Health related Quality of Life (90 day) assessed by Euroqol tool (EQ-5D-5L) | 90 days post ICU discharge
  Health related Quality of Life (90 day) assessed by Euroqol tool (EQ-5D-5L). Scale is between 5-25 which lower scores having the better outcome.
Health related Quality of Life (180 day) assessed by Euroqol tool (EQ-5D-5L) | 180 days post ICU discharge
  Health related Quality of Life (180 day) assessed by Euroqol tool (EQ-5D-5L). Scale is between 5-25 which lower scores having the better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Walsh, MBChB MD MSc, Principal Investigator — University of Edinburgh
Locations (38):
- United Kingdom (38):
  - Belfast Health & Social Care Trust, Belfast
  - South Eastern Health and Social Trust, Belfast
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - North Bristol NHS Trust, Bristol
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff and Vale University Health Board, Cardiff
  - Countess of Chester Hospital NHS Foundation Trust, Chester
  - The Dudley Group NHS Foundation Trust, Dudley
  - NHS Dumfries and Galloway, Dumfries
  - NHS Lothian, Edinburgh
  - Medway NHS Foundation Trust, Gillingham
  - NHS Greater Glasgow and Clyde, Glasgow
  - Harrogate and District NHS Trust, Harrogate
  - Wye Valley NHS Trust, Hereford
  - The Queen Elizabeth Hospital Kings Lynn NHS Foundation Trust, Kings Lynn
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester, Leicester
  - Lewisham and Greenwich NHS Trust, Lewisham
  - Aintree University Hospital Foundation Trust, Liverpool
  - Royal Liverpool and Broadgreen University Hospitals NHS Trust, Liverpool
  - Guys and St Thomas NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Manchester University Foundation Trust, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Aneurin Bevan University Health Board, Newport
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust., Oxford
  - Poole Hospitals NHS Foundation Trust, Poole
  - University Hospital Southampton NHSFT, Southampton
  - North Tees and Hartlepool NHS Foundation Trust, Stockton-on-Tees
  - Taunton and Somerset NHS Foundation Trust, Taunton
  - West Hertfordshire Hospitals NHS Trust, Watford

IPD SHARING:
Plan to Share IPD: Yes
The final trial dataset will be held by the University of Edinburgh on a secure password protected drive. Co-investigators will have the right to access the final data set for the purpose of additional analyses that are consistent with the consent provided by participants. Similarly, any external party can approach the co-investigators to request access to the trial data. In all cases, access to the trial dataset will require approval by a majority of the members of the trial management group and the sponsor (or its delegated representative).
Supporting Information: Study Protocol
Time Frame: Currently unknown
Access Criteria: Currently unspecified

REFERENCES:
- [Derived] Emerson LM, Blackwood B, Kydonaki K, McKenzie C, Walsh TS, Aitken LM. The experiences of bedside nurses delivering an intensive care sedation study: A process evaluation within the A2B trial. J Intensive Care Soc. 2025 Nov 6:17511437251381951. doi: 10.1177/17511437251381951. Online ahead of print. PMID 41220595
- [Derived] Walsh TS, Parker RA, Aitken LM, McKenzie CA, Emerson L, Boyd J, Macdonald A, Beveridge G, Giddings A, Hope D, Irvine S, Tuck S, Lone NI, Kydonaki K, Norrie J, Brealey D, Antcliffe D, Reay M, Williams A, Bewley J, Creagh-Brown B, McAuley DF, Dark P, Wise MP, Gordon AC, Perkins GD, Reade MC, Blackwood B, MacLullich A, Glen R, Page VJ, Weir CJ; A2B Trial Investigators. Dexmedetomidine- or Clonidine-Based Sedation Compared With Propofol in Critically Ill Patients: The A2B Randomized Clinical Trial. JAMA. 2025 Jul 1;334(1):32-45. doi: 10.1001/jama.2025.7200. PMID 40388916
- [Derived] Aitken LM, Emerson LM, Kydonaki K, Blackwood B, Creagh-Brown B, Lone NI, McKenzie CA, Reade MC, Weir CJ, Wise MP, Walsh TS. Alpha 2 agonists for sedation to produce better outcomes from critical illness (A2B trial): protocol for a mixed-methods process evaluation of a randomised controlled trial. BMJ Open. 2024 Apr 5;14(4):e081637. doi: 10.1136/bmjopen-2023-081637. PMID 38580355
- [Derived] Walsh TS, Aitken LM, McKenzie CA, Boyd J, Macdonald A, Giddings A, Hope D, Norrie J, Weir C, Parker RA, Lone NI, Emerson L, Kydonaki K, Creagh-Brown B, Morris S, McAuley DF, Dark P, Wise MP, Gordon AC, Perkins G, Reade M, Blackwood B, MacLullich A, Glen R, Page VJ. Alpha 2 agonists for sedation to produce better outcomes from critical illness (A2B Trial): protocol for a multicentre phase 3 pragmatic clinical and cost-effectiveness randomised trial in the UK. BMJ Open. 2023 Dec 10;13(12):e078645. doi: 10.1136/bmjopen-2023-078645. PMID 38072483

DOCUMENTS (2):
  • Study Protocol (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT03653832/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT03653832/SAP_001.pdf